CLINICAL TRIAL: NCT01935115
Title: A Prospective Randomized Double Blinded Control Trial Using Ketamine or Propofol Anesthesia for Electroconvulsive Therapy: Improving Treatment-Resistant Depression
Brief Title: Comparing Ketamine and Propofol Anesthesia for Electroconvulsive Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatoon Health Region (Other); Royal University Hospital Foundation (Other); Schulman Research Award (Unknown)
Responsible Party: Principal Investigator, Jonathan Gamble, M.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UofSKetamine-01
Record Dates: First submitted 2013-08-26; First posted 2013-09-04 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Treatment Resistant Depression
Keywords: Depression; MDD; Treatment Resistant Depression; Electroconvulsive Therapy; ECT; Ketamine; Propofol; NMDA
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression | interventions — Propofol; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Active Comparator): The control group will receive propofol 1 mg/kg and remifentanil 1 mcg/kg intravenously
  Interventions: Drug: Propofol
- Ketamine (Experimental): Study group will receive ketamine 0.75 mg/kg and remifentanil 1 mcg/kg intravenously
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Propofol — Propofol anesthesia for ECT
  Other Names: Diprivan
  Arms: Propofol
Drug: Ketamine — Ketamine anesthesia for ECT
  Other Names: Ketalar
  Arms: Ketamine

SUMMARY:
To determine the effect of ketamine, compared to propofol, when used an an anesthetic agent for electroconvulsive therapy (ECT) in the treatment of major depressive disorder (MDD). We hypothesize that ketamine, compared to propofol, will improve the the symptoms of MDD when used as the anesthetic agent to facilitate ECT. Additionally, we hypothesize the dissociative and cardiovascular effects of ketamine will be minimal.

DETAILED DESCRIPTION:
Treatment resistant depression is a common and disabling condition. The delayed onset of action and side effects exhibited by oral antidepressants are significant limitations. An alternative and well-established therapy is electroconvulsive therapy (ECT). ECT has rapid antidepressant effect beginning with the completion of the first session. Nevertheless, like oral medications, patients treated with ECT can develop treatment resistance or failure to respond. There is great need for a novel approach to treatment-resistant depression; one that that is safe, has rapid onset, and is sustained.

Pharmaceutical agents with rapid antidepressant effects are a new and promising paradigm in the research for treatment of MDD. A potential therapeutic target is glutamate based signal transmission because glutamate transmission is abnormally regulated in the limbic/cortical areas of many depressed people. Glutamatergic modulating agents, in particular ketamine, have been shown to induce rapid antidepressant effects both in both preclinical models and humans. Additionally, ketamine has been shown to have persistent antidepressive effect.

Presently worldwide, propofol is one of the most commonly used anesthetic agents for ECT. There are 2 main disadvantages to this practice. First, propofol has no antidepressive effect. Second, propofol is a potent anticonvulsant that may worsen the quality of the ECT induced seizures. A recent open-label trial compared ketamine to propofol for anesthesia during ECT and demonstrated a significant improvement of depression in the ketamine arm. Ketamine is routinely used to provide safe general anesthesia as well as procedural sedation, analgesia, and amnesia. The combination of the intrinsic antidepressant effects of ketamine with electroconvulsive therapy is a promising concept in clinical research.

This study will include planned interim analysis to ensure patients safety. This analysis will be performed by a statistician who is blinded to group allocation after 20 and after 40 patients. An independent safety committee will informed of the results of the interim analysis including side effects and complications and will have the option to adjust the drug dosage or to discontinue the trial.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the diagnostic criteria for major depression according to the Diagnostic and Statistical Manual of Mental Disorders (most recent edition)
* Failure to respond to at least 2 adequate drug therapies for the current depression episode
* MADRS score of 20 or above (moderate - severe
* ASA physical status classification I to III

Exclusion Criteria:

* Inability to obtain informed consent
* ASA physical status classification IV
* Complication by any serious physical diseases such as cardiovascular disease (including untreated HTN), respiratory disease, cerebrovascular disease, intracranial HTN (including glaucoma), or seizures
* Presence of foreign body (including pacemaker)
* Pregnancy
* Allergies to anesthetics used in study Includes: a) Ketamine b) Propofol c) Eggs d) Egg products e) Soybeans f) Soy products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome is defined as the number of ECT treatments required to reach a 50% reduction in baseline MADRS (Montgomery-Asberg Depression Scale) score. | After 8 treatments or completion of therapy for an expected average of 4 weeks
  Standard of care for ECT in the Saskatoon Health Region are biweekly sessions for a total of 8 treatments. Occasionally, a patient meets early remission and may not require the full 8 treatments and may be eligible for early withdrawal.

SECONDARY OUTCOMES:
Change in CADSS (Clinician Administered Dissociative States Scale) | 30 minutes after each ECT session and one day after each ECT session for an expected average of 4 weeks
  The CADSS is used to assess states of clinical dissociation; a potential side effect of ketamine. A baseline CADSS will be obtained one day prior to start of ECT. Additional scores will be assessed 30 minutes after each therapy as well as one day post-therapy on the ward.
Change in ALS-18 (Affective Lability Scale) | 30 days after final ECT session for an expected average duration of 2 months
  A baseline ALS-18 score will be obtained. 30 days after completion of therapy, another score will be collected.
Change in ECT energy settings and seizure quality | Within 30 minutes of each treatment for an expected average of 4 weeks
  We will document energy settings used by the psychiatrist as well as duration and quality of seizures achieved.
Hemodynamic instability and respiratory complications | 1 hour after each ECT for an expected average of 4 weeks
  Any hemodynamic or respiratory instability requiring unanticipated intervention will be recorded as well as the treatment for the event recorded. Type of intervention will also be documented.
Time to discharge | 1 hour after each treatment for an expected average of 4 weeks
  Total time spend in the post-anesthetic recovery unit will be recorded.
Change in MADRS score | 24 hours after each treatment and 30 days after final treatment for an expected average of 2 months
  A baseline MADRS score will be conducted one day prior to ECT. Additional scores will be obtained one day after each ECT session. A final MADRS score will be assessed 30 days after completion of ECT.
The number of ECT sessions required to achieve depression remission (MADRS ≤10) | Number of ECT treatments to achieve depression remission (MADRS) or completion of therapy up to 4 weeks
  Standard of care for ECT in the Saskatoon Health Region are biweekly sessions for a total of 8 treatments. Occasionally, a patient meets early remission and may not require the full 8 treatments and may be eligible for early withdrawal.
The proportion of depressed patients (MADRS > 20) at 30 days after the last ECT session | 30 days after the last ECT session, up to 60 days after ECT initiation.
  The proportion of patients in each group who have severe depression 30 days after their last ECT session. This is a measure of longer term efficacy of treatment effect.
Change in systolic blood pressure | During ECT, up to 8 treatments or 4 weeks
  Increases or decreases in baseline systolic blood pressure at any point during the anesthetic care will be categorically recorded as minimal change (20 - 50 mm Hg from baseline) and significant change (more than 50 mm Hg from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gamble, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Zarate CA Jr, Brutsche NE, Ibrahim L, Franco-Chaves J, Diazgranados N, Cravchik A, Selter J, Marquardt CA, Liberty V, Luckenbaugh DA. Replication of ketamine's antidepressant efficacy in bipolar depression: a randomized controlled add-on trial. Biol Psychiatry. 2012 Jun 1;71(11):939-46. doi: 10.1016/j.biopsych.2011.12.010. Epub 2012 Jan 31. PMID 22297150
- [Background] Diazgranados N, Ibrahim L, Brutsche NE, Newberg A, Kronstein P, Khalife S, Kammerer WA, Quezado Z, Luckenbaugh DA, Salvadore G, Machado-Vieira R, Manji HK, Zarate CA Jr. A randomized add-on trial of an N-methyl-D-aspartate antagonist in treatment-resistant bipolar depression. Arch Gen Psychiatry. 2010 Aug;67(8):793-802. doi: 10.1001/archgenpsychiatry.2010.90. PMID 20679587
- [Background] Okamoto N, Nakai T, Sakamoto K, Nagafusa Y, Higuchi T, Nishikawa T. Rapid antidepressant effect of ketamine anesthesia during electroconvulsive therapy of treatment-resistant depression: comparing ketamine and propofol anesthesia. J ECT. 2010 Sep;26(3):223-7. doi: 10.1097/YCT.0b013e3181c3b0aa. PMID 19935085
- [Background] Wang X, Chen Y, Zhou X, Liu F, Zhang T, Zhang C. Effects of propofol and ketamine as combined anesthesia for electroconvulsive therapy in patients with depressive disorder. J ECT. 2012 Jun;28(2):128-32. doi: 10.1097/YCT.0b013e31824d1d02. PMID 22622291
- [Derived] Gamble JJ, Bi H, Bowen R, Weisgerber G, Sanjanwala R, Prasad R, Balbuena L. Ketamine-based anesthesia improves electroconvulsive therapy outcomes: a randomized-controlled study. Can J Anaesth. 2018 Jun;65(6):636-646. doi: 10.1007/s12630-018-1088-0. Epub 2018 Feb 21. PMID 29700801